CLINICAL TRIAL: NCT02823145
Title: An Open-Label Extension Trial to Assess the Long-Term Safety of ZX008 (Fenfluramine Hydrochloride HCl) Oral Solution as an Adjunctive Therapy in Children and Young Adults With Dravet Syndrome
Brief Title: An Open-Label Extension Trial to Assess the Long-Term Safety of ZX008 (Fenfluramine Hydrochloride HCl) Oral Solution in Children and Young Adults With Dravet Syndrome
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Zogenix International Limited, Inc., a subsidiary of Zogenix, Inc. (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZX008-1503; 2016-002804-14 (EudraCT Number)
Record Dates: First submitted 2016-06-13; First posted 2016-07-06 (Estimated); Results first posted 2023-09-25 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Dravet Syndrome
Keywords: seizure; tonic clonic; epilepsy; myoclonic; encephalopathy
MeSH Terms: conditions — Epilepsies, Myoclonic; Seizures; Epilepsy; Brain Diseases | interventions — Fenfluramine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- ZX008 (Experimental): ZX008 is supplied as an oral solution in a concentration of 2.5 mg/mL. Subjects will be titrated to an effective dose beginning with 0.2 mg/kg/day (maximum: 30 mg/day).
  Interventions: Drug: ZX008 (Fenfluramine Hydrochloride)

INTERVENTIONS:
Drug: ZX008 (Fenfluramine Hydrochloride)

SUMMARY:
This is an international, multicenter, open-label, long-term safety study of ZX008 in subjects with Dravet syndrome.

DETAILED DESCRIPTION:
This is an international, multicenter, open-label, long-term safety study of ZX008 in pediatric and young adult subjects with Dravet syndrome who participated in one of the core studies (ZX008-1501 and ZX008-1502) and are candidates for continuous treatment for an extended period of time. This trial will consist of a 36-month Open-Label Extension (OLE) Treatment Period and a 2-week Post-Dosing Period.

ELIGIBILITY:
Key Inclusion Criteria:

* Male or non-pregnant, non-lactating female, age 2 to 18 years, inclusive as of the day of the core study Screening Visit.
* Satisfactory completion of the core study in the opinion of the investigator and the sponsor.
* Subjects who are >18 to ≤35 years of age at the time of screening and did not participate in one of the core studies may be eligible for participation.
* A documented medical history to support a clinical diagnosis of Dravet syndrome, where convulsive seizures are not completely controlled by current antiepileptic drugs.
* Parent/caregiver is willing and able to be compliant with diary completion, visit schedule and study drug accountability.
* Subject's parent/caregiver has been compliant with diary completion during the core study, in the opinion of the investigator (eg, at least 90% compliant).

Key Exclusion Criteria:

* Current or past history of cardiovascular or cerebrovascular disease, myocardial infarction or stroke.
* Current cardiac valvulopathy or pulmonary hypertension that is clinically significant and warrants discontinuation of study medication.
* Current or past history of glaucoma.
* Moderate or severe hepatic impairment.
* Receiving concomitant therapy with: centrally-acting anorectic agents; monoamineoxidase inhibitors; any centrally-acting compound with clinically appreciable amount of serotonin agonist or antagonist properties, including serotonin reuptake inhibition; atomoxetine, or other centrally-acting noradrenergic agonist; cyproheptadine, and/or cytochrome P450 (CYP) 2D6/3A4/2B6 inhibitors/substrates.
* Currently taking carbamazepine, oxcarbamazepine, eslicarbazepine, phenobarbital, or phenytoin, or has taken any of these within the past 30 days, as maintenance therapy.
* A clinically significant condition, or has had clinically relevant symptoms or a clinically significant illness at Visit 1, other than epilepsy, that would negatively impact study participation, collection of study data, or pose a risk to the subject.

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 375 (Actual)
Dates: Start 2016-06-08 (Actual); Primary Completion 2023-01-27 (Actual); Study Completion 2023-01-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Cares, Study Director — 001 844 599 2273
Locations (67):
- United States (24):
  - Phoenix Children's Hospital, Phoenix, Arizona
  - Center for Neurosciences - Tucson, Tucson, Arizona
  - Children's Hospital of Orange County, Orange, California
  - Rady Children's Hospital San Diego, San Diego, California
  - University of California San Francisco, San Francisco, California
  - The Children's Hospital Colorado, Aurora, Colorado
  - NW FL Clinical Research Group, LLC, Gulf Breeze, Florida
  - Miami Children's Hospital Brain Institute, Miami, Florida
  - Neurology and Epilepsy Research Center, Orlando, Florida
  - Clinical Integrative Research Center of Atlanta, Panda Neurology, Atlanta, Georgia
  - Ann and Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois
  - Massachusetts General Hospital, Boston, Massachusetts
  - Boston Children's Hospital, Boston, Massachusetts
  - Children's Hospital Of Michigan, Detroit, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Minnesota Epilepsy Group, P.A., Saint Paul, Minnesota
  - Institute of Neurology and Neurosurgery at St. Barnabus, Livingston, New Jersey
  - University Hospitals Cleveland Medical Center, Cleveland, Ohio
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Le Bonheur Children's Hospital, Memphis, Tennessee
  - Cook Children's Medical Center, Fort Worth, Texas
  - University of Utah, Salt Lake City, Utah
  - Seattle Children's Hospital, Seattle, Washington
  - MultiCare Institute for Research & Innovation, Tacoma, Washington
- Australia (3):
  - Melbourne Brain Centre Austin Hospital, Heidelberg
  - Children's Health Queensland Hospital and Health Service at Lady Cilento Children's Hospital, South Brisbane
  - The Children's Hospital Westmead Dept. of Neurology and Neurosurgery, Westmead
- Universitair Ziekenhuis Antwerpen, Edegem, Belgium
- Canada (2):
  - Centre Hospitalier Universitaire Sainte-Justine, Montreal
  - British Columbia Children's Hospital, Vancouver
- Danish National Epilepsy Centre, Dianalund, Denmark
- France (6):
  - CHU Amiens-Picardie Service De Neurologie Pediatrique, Amiens
  - CHU De Bordeaux Service De Pédiatrie Médicale, Bordeaux
  - CHRU Lille Antenne Pédiatrique Du CIC - Hôpital Jeanne De Flandre, Lille
  - HOPITAL DEL LA TIMONE - HOPITAL HENRI GASTAUT Hôpital De La Timone Neurologie Pédiatrique Pneumologie Pédiatrique Et Médecine Infantile, Marseille
  - Hôpital Robert Debré Pôle: Pédiatrie Médicale Service: Neurologie Et Maladies Métaboliques, Paris
  - Hôpital Universitaire Necker-Enfants Malades Service de neurologie pédiatrique Centre de référence épilepsies rares (CReER), Paris
- Germany (8):
  - DRK Kliniken Berlin - Westend Epilepsiezentrum / Neuropaediatrie, Berlin
  - Krankenhaus Mara Epilepsie-Zentrum Bethel, Bielefeld
  - Universitaetsklinikum Freiburg Zentrum fuer Kinder- und Jugendmedizin, Freiburg im Breisgau
  - Universitaetsklinikum Jena Klinik fuer Kinder- und Jugendmedizin Neuropaediatrie, Jena
  - Universitaetsklinikum Schleswig-Holstein Campus Kiel Klinik fuer Neuropaediatrie, Kiel
  - Kleinwachau Saechsisches Epilepsiezentrum Radeberg gemeinnuetzige GmbH, Radeberg
  - Universitaetsklinik fuer Kinder- und Jugendmedizin Abteilung III, Tübingen
  - Schoen Klinik Vogtareuth Neuropaediatrie und Neurologische Rehabilitation, Epilepsiezentrum fuer Kinder und Jugendlische, Tagesklinik fuer Neuropaediatrie, Vogtareuth
- Italy (8):
  - AOU Anna Meyer Clinica di Neurologia Pediatrica, Florence
  - Istituto Pediatrico Giannina Gaslini Dipartimento di Neurologia, Genova
  - A.O. Carlo Poma, Mantova
  - Istituto Neurologica Carlo Besta, Milan
  - Ospedale Fatebenefratelli e Oftalmico, Milan
  - Policlinico A. Gemelli, Roma
  - U.O. Neurologia Dipartimento di Neuroscienze Ospedale Pediatrico Bambino Gesù, Roma
  - Ospedale Civile Maggiore di Borgo Trento - Ospedale della Donna e del Bambino, Verona
- Japan (3):
  - Saitama Children's Medical Center, Saitama
  - National Epilepsy Center Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka
  - Tokyo Women's Medical University Hospital, Tokyo
- Netherlands (2):
  - Kempenhaeghe, Heeze
  - Stichting Epilepsie Instellingen Nederland, Zwolle
- Spain (3):
  - Hospital Sant Joan de Déu, Barcelona
  - Hospital Ruber Internacional Primera Planta Servicio de Neurologia, Madrid
  - Clinica Universitaria de Navarra Fase 4. Segunda planta, Consulta de Pediatria, Pamplona
- United Kingdom (6):
  - Birmingham Children Hospital NHS Foundation Trust, Birmingham
  - Institute of Neurosciences Queen Elizabeth University Hospital, Glasgow
  - Alder Hey Hospital, Liverpool
  - Great Ormond Street Hospital for Children NHS Foundation Trust, London
  - St. Thomas Hospital, London
  - Sheffield Children's Hospital, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe, or global development is discontinued, and 18 months after trial completion. Investigators may request access to anonymized individual patient-level data and redacted trial documents which may include: analysis-ready datasets, study protocol, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a prespecified time, typically 12 months, on a password protected portal. This plan may change if the risk of re-identifying trial participants is determined to be too high after the trial is completed; in this case and to protect participants, individual patient-level data would not be made available.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data from this trial may be requested by qualified researchers six months after product approval in the US and/or Europe or global development is discontinued, and 18 months after trial completion.
Access Criteria: Qualified researchers may request access to anonymized IPD and redacted study documents which may include: raw datasets, analysis-ready datasets, study protocol, blank case report form, annotated case report form, statistical analysis plan, dataset specifications, and clinical study report. Prior to use of the data, proposals need to be approved by an independent review panel at www.Vivli.org and a signed data sharing agreement will need to be executed. All documents are available in English only, for a pre-specified time, typically 12 months, on a password protected portal.
URL: https://www.Vivli.org

REFERENCES:
- [Result] Scheffer IE, Nabbout R, Lagae L, Devinsky O, Auvin S, Thiele EA, Wirrell EC, Polster T, Specchio N, Pringsheim M, Imai K, Lock MD, Langlois M, Roper RZ, Lothe A, Sullivan J. Long-term safety and effectiveness of fenfluramine in children and adults with Dravet syndrome. Epilepsia. 2025 Jun;66(6):1919-1932. doi: 10.1111/epi.18342. Epub 2025 Mar 12. PMID 40072476
- [Derived] Cross JH, Galer BS, Gil-Nagel A, Devinsky O, Ceulemans B, Lagae L, Schoonjans AS, Donner E, Wirrell E, Kothare S, Agarwal A, Lock M, Gammaitoni AR. Impact of fenfluramine on the expected SUDEP mortality rates in patients with Dravet syndrome. Seizure. 2021 Dec;93:154-159. doi: 10.1016/j.seizure.2021.10.024. Epub 2021 Nov 2. PMID 34768178

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study started to enroll participants in Jun 2016 and concluded in Jan 2023. Participants who completed 14 weeks treatment in any of the core studies ZX008-1501/ZX008-1502 (NCT02682927), or ZX008-1504 (NCT02926898) Cohort 2, or completed ZX008-1504 Cohort 1 study, and de novo participants were eligible to participate in this study.
Pre-assignment Details: The Participant Flow refers to the Safety (SAF) Population.
Groups:
- Not Treated: Participant (de novo) signed the informed consent form (ICF) but never received any study medication during the study.
- Any ZX008 Open Label Dose: Participants received ZX008 0.2 milligram per kilogram per day (mg/kg/day) as an oral solution, twice a day (bid), in equally divided doses with food for 1 month. After 1 month, investigator might have adjusted the dose of each participant based on effectiveness and tolerability. Participants who were not receiving concomitant stiripentol, dose changes should be made in increments of 0.2 mg/kg/day, to a maximum of 0.8 mg/kg/day but not to exceed total dose of 30 mg/day for 42 months of OLE Period. Participants who were receiving concomitant stiripentol, the first dose change was 0.4 mg/kg/day and the final dose change was to 0.5 mg/kg/day, but not to exceed 20 mg/day for 42 months of OLE Period.
Period: Enrollment
Arm/Group | Not Treated | Any ZX008 Open Label Dose
Started | 1 | 374
Completed | 0 | 374
Not Completed | 1 | 0
Not completed — Other | 1 | 0
Period: Treatment
Arm/Group | Not Treated | Any ZX008 Open Label Dose
Started | 0 | 374
Completed | 0 | 49
Not Completed | 0 | 325
Not completed — Adverse Event | 0 | 11
Not completed — Death | 0 | 3
Not completed — Family Decision | 0 | 1
Not completed — IP approved and subject moved to commercial drug | 0 | 1
Not completed — Lack of Efficacy | 0 | 48
Not completed — Non-Compliance With E-Diary | 0 | 1
Not completed — Physician Decision | 0 | 2
Not completed — Subject has transitioned to study 1900 OLE study | 0 | 225
Not completed — Subject needed to take prohibited medication | 0 | 1
Not completed — Subject transferred to direct access programme | 0 | 1
Not completed — Switching to commercially available drug | 0 | 11
Not completed — Transitioned to commercial supply of medication | 0 | 1
Not completed — Withdrawal By Caregiver | 0 | 1
Not completed — Withdrawal by sponsor due to lack of compliance | 0 | 1
Not completed — Withdrawal by Subject | 0 | 16
Not completed — Reason unknown | 0 | 1

BASELINE CHARACTERISTICS:
Population: Baseline characteristics refers to the Safety (SAF) population which included all enrolled participants who received at least one dose of ZX008 during the open label extension (OLE). As pre-specified in the SAP, participant Demographics and Baseline Characteristics were summarized for the safety population.
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 374
Age, Continuous [Mean (Standard Deviation); unit: years] | 10.3 (6.12)
Age, Customized [Count of Participants; unit: Participants]
  <6 years | 92
  6-18 years | 250
  >18 years | 32
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 172
  Male | 202
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 275
  Black or African American | 5
  Asian | 31
  American Indian or Alaska Native | 2
  Other | 17
  Not Reported | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 44
  Not Hispanic or Latino | 267
  Not Reported | 55
  Unknown | 8

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) During the Open-label Extension (OLE) Treatment Period
Description: Treatment-emergent adverse events (TEAE) were defined as any AEs that based on start date information occurs after the first intake of study treatment.
Time Frame: From Day 1 to End of OLE Treatment Period - End of Study (EOS) Visit (Month 42)
Population: Safety (SAF) population included all enrolled participants who received at least one dose of ZX008 during the OLE.
Measure: Number; unit: percentage of participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 374
percentage of participants | 98.1

2. Primary Outcome: Percentage of Participants With Treatment-emergent Adverse Events (TEAEs) Leading to Withdrawal From Investigational Medicinal Product (IMP) During the OLE Treatment Period
Description: A TEAE was defined as any AE that based on start date information occurs after the first intake of study treatment. Percentage of participants with TEAEs leading to withdrawal from IMP during OLE Treatment Period were reported.
Time Frame: From Day 1 to End of OLE Treatment Period - EOS Visit (Month 42)
Population: Safety (SAF) population included all enrolled participants who received at least one dose of ZX008 during the OLE.
Measure: Number; unit: percentage of participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 374
percentage of participants | 3.5

3. Primary Outcome: Percentage of Participants With Serious Treatment-emergent Adverse Events (TEAEs) During the OLE Treatment Period
Description: Serious Adverse event (SAE) was defined as any untoward medical occurrence that at any dose: • results in death, • is life-threatening threatening, • results in initial inpatient hospitalization or prolongation of hospitalization, •results in persistent or significant disability or incapacity, • results in a congenital anomaly/birth defect, • results in any medically significant event that did not meet any of the other 5 SAE criteria, but which was judged by a physician to potentially jeopardize the participant or require medical or surgical intervention to prevent one of the above outcomes listed as an SAE criterion.
Time Frame: From Day 1 to End of OLE Treatment Period - EOS Visit (Month 42)
Population: Safety (SAF) population included all enrolled participants who received at least one dose of ZX008 during the OLE.
Measure: Number; unit: percentage of participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 374
percentage of participants | 26.5

4. Secondary Outcome: Change From Baseline (Core) in Convulsive Seizure Frequency Per 28 Days From Day 1 to End of Study (EOS) Visit (Month 42) in the OLE Treatment Period
Description: Baseline (Core) was defined as Baseline prior to double-blind treatment in the core studies (ZX008-1501/ZX008-1502, and ZX008-1504 Cohort 2). Participants in 1504- Cohort 1 and de novo participants (who entered 1503 without having been in any of the core studies) did not have a Baseline (Core), and were not included in the analysis of this outcome measure. The total number of convulsive seizures from Day 1 to EOS was divided by the total number of days from Day 1 to EOS with nonmissing diary data and the result was then multiplied by 28 to get a 28-day convulsive seizure frequency (CSF). The change from Baseline for any individual participant was calculated by subtracting the Baseline (Core) from the post-baseline value. Monthly (28 day) CSF was based on electronic diary data obtained for each participant.
Time Frame: From Day 1 to End of OLE Treatment Period (EOS Visit - up to Month 42), compared to Baseline (Core)
Population: Modified Intent-to-Treat (mITT) population included all enrolled participants who received at least one dose of ZX008 and had at least 1 month of valid seizure data during the OLE.
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 324
seizure frequency per 28 days | -6.67 [-1757.8 to 751.3]

5. Secondary Outcome: Change From Baseline (Core) in Convulsive Seizure Frequency Per 28 Days From Month 2 to EOS (Month 42) in the OLE Treatment Period
Description: Baseline (Core) was defined as Baseline prior to double-blind treatment in the core studies. Participants in 1504-Cohort 1 and de novo participants did not have a Baseline (Core), and were not included in the analysis of this outcome measure. The total number of convulsive seizures from Month 2 to EOS was divided by the total number of days from Month 2 to EOS with nonmissing diary data and the result was then multiplied by 28 to get a 28-day CSF. The change from Baseline for any individual participant was calculated by subtracting the Baseline (Core) from the post-baseline value. Monthly (28 day) CSF was based on electronic diary data obtained for each participant.
Time Frame: From Month 2 to End of OLE Treatment Period (EOS Visit - up to Month 42), compared to Baseline (Core)
Population: mITT population included all enrolled participants who received at least one dose of ZX008 and had at least 1 month of valid seizure data during the OLE. Here, number of participants analyzed included those participants who were evaluable for the assessment.
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 323
seizure frequency per 28 days | -7.04 [-1986.9 to 816.4]

6. Secondary Outcome: Convulsive Seizure Frequency (CSF) Per 28 Days During the OLE Treatment Period (to Month 36)
Description: Monthly (28 day) CSF was based on electronic diary data obtained for each participant. The total number of convulsive seizures in the ith interval (CSF in OLE, where, i=1, 2, 3, … , 14 ) was divided by the total number of days in the ith interval with nonmissing diary data and the result was then multiplied by 28 to get a 28-day CSF of OLE.
Time Frame: At Month 1, Month 2, Month 3, Month 4-6, Month 7-9, Month 10-12, Month 13-15, Month 16-18, Month 19-21, Month 22-24, Month 25-27, Month 28-30, Month 31-33, and Month 34-36
Population: mITT population included all enrolled participants who received at least one dose of ZX008 and had at least 1 month of valid seizure data during the OLE. Here, number analyzed signifies participants who were evaluable at specified time points.
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 324
seizure frequency per 28 days
  Month 1 | 6.53 [0.0 to 4876.9]
  Month 2: number analyzed (Participants) | 323
  Month 2 | 4.67 [0.0 to 3392.7]
  Month 3: number analyzed (Participants) | 320
  Month 3 | 4.67 [0.0 to 2593.7]
  Month 4-6: number analyzed (Participants) | 316
  Month 4-6 | 4.36 [0.0 to 1725.5]
  Month 7-9: number analyzed (Participants) | 299
  Month 7-9 | 3.82 [0.0 to 310.8]
  Month 10-12: number analyzed (Participants) | 284
  Month 10-12 | 4.04 [0.0 to 362.4]
  Month 13-15: number analyzed (Participants) | 280
  Month 13-15 | 3.11 [0.0 to 215.0]
  Month 16-18: number analyzed (Participants) | 262
  Month 16-18 | 3.42 [0.0 to 243.3]
  Month 19-21: number analyzed (Participants) | 247
  Month 19-21 | 3.42 [0.0 to 372.4]
  Month 22-24: number analyzed (Participants) | 234
  Month 22-24 | 2.80 [0.0 to 489.5]
  Month 25-27: number analyzed (Participants) | 187
  Month 25-27 | 2.80 [0.0 to 747.3]
  Month 28-30: number analyzed (Participants) | 151
  Month 28-30 | 2.80 [0.0 to 242.5]
  Month 31-33: number analyzed (Participants) | 116
  Month 31-33 | 3.21 [0.0 to 224.0]
  Month 34-36: number analyzed (Participants) | 73
  Month 34-36 | 2.74 [0.0 to 56.0]

7. Secondary Outcome: Convulsive Seizure Frequency (CSF) by Mean Daily Dose During the Overall OLE Treatment Period
Description: Convulsive seizure frequency over time, reported as per 28 days was analyzed by the actual dose administered. Participants were grouped into low (0.2 to <0.4 mg/kg), medium (0.4 to <0.6 mg/kg), and high dose (>0.6 mg/kg) groups depending on their mean daily doses of ZX008 during the OLE Treatment period. For each participant, the seizure frequency per 28 days was calculated as the number of seizures recorded during the period, divided by the number of days in the period and multiplied by 28. The convulsive seizure frequency was calculated from all available data collected.
Time Frame: From Day 1 to End of OLE Treatment Period - End of Study (EOS) Visit (Month 42)
Population: mITT population included all enrolled participants who received at least one dose of ZX008 and had at least 1 month of valid seizure data during the OLE. Here, number analyzed represents the number of participants categorized by mean daily dose.
Measure: Median (Full Range); unit: seizure frequency per 28 days
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 324
seizure frequency per 28 days
  ZX008 Low Dose (0 - <0.4 mg/kg/day): number analyzed (Participants) | 90
  ZX008 Low Dose (0 - <0.4 mg/kg/day) | 3.94 [0.0 to 2215.3]
  ZX008 Medium Dose (0.4 - <0.6 mg/kg/day): number analyzed (Participants) | 113
  ZX008 Medium Dose (0.4 - <0.6 mg/kg/day) | 4.80 [0.0 to 113.6]
  ZX008 High Dose (>=0.6 mg/kg/day): number analyzed (Participants) | 121
  ZX008 High Dose (>=0.6 mg/kg/day) | 6.00 [0.1 to 942.8]

8. Secondary Outcome: Percentage of Participants With Changes in Antiepileptic Drug (AED) Medications During First 6 Months of OLE Treatment Period
Description: Participants in the study were required to be on stable background therapy for the first 6 months of treatment, after which background AEDs could be reduced or withdrawn so long as one background AED remained. The percentage of participants who had changes in dose or type of concomitant AED medications during the first, second, third, fourth, fifth, and sixth months were analyzed and reported.
Time Frame: At Month 1, 2, 3, 4 , 5, and 6 of OLE Treatment Period
Population: mITT population included all enrolled participants who received at least one dose of ZX008 and had at least 1 month of valid seizure data during the OLE.
Measure: Number; unit: percentage of participants
Arm/Group | Any ZX008 Open Label Dose
Number analyzed (Participants) | 324
percentage of participants
  OLE Month 1 | 5.2
  OLE Month 2 | 7.1
  OLE Month 3 | 7.4
  OLE Month 4 | 8.3
  OLE Month 5 | 6.8
  OLE Month 6 | 9.6

ADVERSE EVENTS:
Time Frame: From Day 1 up to 42 months
Description: A TEAE was defined as any AE that based on start date information occurs after the first intake of study treatment. The Safety (SAF) population was the set of all enrolled subjects who received at least one dose of ZX008 during the OLE. As pre-specified in the SAP, safety analyses were performed on the SAF Population.
Arm/Group | Any ZX008 Open Label Dose
All-Cause Mortality (participants affected / at risk) | 3/374
Serious Adverse Events (participants affected / at risk) | 99/374
Other Adverse Events (participants affected / at risk) | 342/374
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Any ZX008 Open Label Dose (N=374)
Atrioventricular block second degree (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 2 (2)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Duodenal perforation (Gastrointestinal disorders) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 2 (2)
Enterovesical fistula (Gastrointestinal disorders) | 1 (1)
Haematemesis (Gastrointestinal disorders) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 1 (1)
Tooth disorder (Gastrointestinal disorders) | 1 (1)
Abasia (General disorders) | 1 (1)
Fatigue (General disorders) | 1 (1)
Hypothermia (General disorders) | 1 (1)
Impaired healing (General disorders) | 1 (1)
Sudden unexplained death in epilepsy (General disorders) | 3 (3)
Atypical pneumonia (Infections and infestations) | 1 (1)
Bronchitis (Infections and infestations) | 1 (1)
Bronchitis viral (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 2 (2)
Enterovirus infection (Infections and infestations) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1)
Epstein-Barr virus infection (Infections and infestations) | 1 (1)
Gastroenteritis (Infections and infestations) | 3 (3)
Gastroenteritis viral (Infections and infestations) | 1 (1)
Helicobacter infection (Infections and infestations) | 1 (1)
Infectious mononucleosis (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 7 (8)
Lower respiratory tract infection (Infections and infestations) | 3 (3)
Lung infection (Infections and infestations) | 1 (1)
Otitis media acute (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 12 (15)
Postoperative wound infection (Infections and infestations) | 2 (2)
Respiratory syncytial virus infection (Infections and infestations) | 1 (1)
Rhinovirus infection (Infections and infestations) | 1 (2)
Sepsis (Infections and infestations) | 3 (4)
Tonsillitis (Infections and infestations) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Varicella (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 5 (5)
Viral pharyngitis (Infections and infestations) | 1 (1)
Viral upper respiratory tract infection (Infections and infestations) | 1 (1)
Abdominal injury (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 1 (1)
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 1 (1)
Concussion (Injury, poisoning and procedural complications) | 1 (1)
Drug dose omission (Injury, poisoning and procedural complications) | 1 (1)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Foreign body aspiration (Injury, poisoning and procedural complications) | 1 (1)
Hand fracture (Injury, poisoning and procedural complications) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 2 (2)
Lower limb fracture (Injury, poisoning and procedural complications) | 1 (1)
Near drowning (Injury, poisoning and procedural complications) | 1 (1)
Blood glucose decreased (Investigations) | 1 (1)
Heart rate decreased (Investigations) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (3)
Feeding intolerance (Metabolism and nutrition disorders) | 1 (1)
Hyperammonaemia (Metabolism and nutrition disorders) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 1 (2)
Aneurysmal bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 1 (1)
Change in seizure presentation (Nervous system disorders) | 5 (6)
Dystonia (Nervous system disorders) | 1 (1)
Encephalopathy (Nervous system disorders) | 1 (1)
Epilepsy (Nervous system disorders) | 1 (1)
Febrile convulsion (Nervous system disorders) | 2 (2)
Generalised tonic-clonic seizure (Nervous system disorders) | 2 (4)
Hyperkinesia (Nervous system disorders) | 2 (2)
Hypotonia (Nervous system disorders) | 1 (1)
Lethargy (Nervous system disorders) | 1 (1)
Movement disorder (Nervous system disorders) | 2 (2)
Myoclonus (Nervous system disorders) | 1 (1)
Petit mal epilepsy (Nervous system disorders) | 1 (1)
Seizure (Nervous system disorders) | 21 (26)
Seizure cluster (Nervous system disorders) | 6 (9)
Status epilepticus (Nervous system disorders) | 15 (18)
Acute psychosis (Psychiatric disorders) | 1 (4)
Agitation (Psychiatric disorders) | 1 (1)
Apathy (Psychiatric disorders) | 1 (1)
Insomnia (Psychiatric disorders) | 3 (3)
Tic (Psychiatric disorders) | 1 (1)
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Apnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 1 (1)
Labial frenectomy (Surgical and medical procedures) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Any ZX008 Open Label Dose (N=374)
Constipation (Gastrointestinal disorders) | 23 (34)
Diarrhoea (Gastrointestinal disorders) | 73 (102)
Vomiting (Gastrointestinal disorders) | 39 (50)
Fatigue (General disorders) | 34 (49)
Pyrexia (General disorders) | 112 (229)
Ear infection (Infections and infestations) | 39 (56)
Gastroenteritis (Infections and infestations) | 32 (34)
Gastroenteritis viral (Infections and infestations) | 20 (21)
Influenza (Infections and infestations) | 45 (50)
Nasopharyngitis (Infections and infestations) | 104 (224)
Rhinitis (Infections and infestations) | 32 (62)
Upper respiratory tract infection (Infections and infestations) | 65 (117)
Viral infection (Infections and infestations) | 27 (40)
Viral upper respiratory tract infection (Infections and infestations) | 19 (36)
Fall (Injury, poisoning and procedural complications) | 25 (26)
Blood glucose decreased (Investigations) | 88 (115)
Echocardiogram abnormal (Investigations) | 67 (82)
Weight decreased (Investigations) | 31 (33)
Decreased appetite (Metabolism and nutrition disorders) | 100 (112)
Hypoglycaemia (Metabolism and nutrition disorders) | 32 (35)
Seizure (Nervous system disorders) | 46 (60)
Somnolence (Nervous system disorders) | 35 (38)
Tremor (Nervous system disorders) | 21 (24)
Abnormal behaviour (Psychiatric disorders) | 22 (28)
Irritability (Psychiatric disorders) | 19 (23)
Cough (Respiratory, thoracic and mediastinal disorders) | 34 (55)
Rash (Skin and subcutaneous tissue disorders) | 20 (20)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2020-08-03): https://cdn.clinicaltrials.gov/large-docs/45/NCT02823145/Prot_000.pdf
  • Statistical Analysis Plan (2020-08-04): https://cdn.clinicaltrials.gov/large-docs/45/NCT02823145/SAP_001.pdf